CLINICAL TRIAL: NCT04066257
Title: An Open-Label, Randomized, Crossover Study to Evaluate the Pharmacokinetic Interaction After Multiple Oral Doses of Tegoprazan, Metronidazole, Tetracycline and Bismuth in Healthy Volunteers
Brief Title: Evaluate the PK of Multiple Oral Doses of Tegoprazan, Metronidazole, Tetracycline and Bismuth in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_111
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Drug-Drug interaction; pharmacokinetic
MeSH Terms: interventions — tegoprazan; Metronidazole; Tetracycline; Bismuth; bismuth tripotassium dicitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50 mg (Active Comparator): Oral administration of Tegoprazan 50 mg twice daily for 7 days
  Interventions: Drug: Tegoprazan
- Tegoprazan 50 mg+MTN 500 mg+TCL 500 mg+BIS 300 mg (Active Comparator): Oral administration of Tegoprazan 50 mg twice daily, Metronidazole 500 mg three times daily, and Tetracycline hydrochloride 500 mg & Tripotassium bismuth dicitrate 300 mg four times daily for 7 days
  Interventions: Drug: Tegoprazan; Drug: Metronidazole; Drug: Tetracycline; Drug: Bismuth
- MTN 500 mg+TCL 500 mg+BIS 300 mg (Active Comparator): Oral administration of Metronidazole 500 mg twice daily, Tetracycline hydrochloride 500 mg & Tripotassium bismuth dicitrate 300 mg four times daily for 7 days
  Interventions: Drug: Metronidazole; Drug: Tetracycline; Drug: Bismuth

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Tegoprazan 50 mg; Tegoprazan 50 mg+MTN 500 mg+TCL 500 mg+BIS 300 mg
Drug: Metronidazole — Metronidazole 250 mg tablet
  Other Names: Flasinyl
  Arms: MTN 500 mg+TCL 500 mg+BIS 300 mg; Tegoprazan 50 mg+MTN 500 mg+TCL 500 mg+BIS 300 mg
Drug: Tetracycline — Tetracycline hydrochloride 250 mg capsule
  Other Names: Teracyclin
  Arms: MTN 500 mg+TCL 500 mg+BIS 300 mg; Tegoprazan 50 mg+MTN 500 mg+TCL 500 mg+BIS 300 mg
Drug: Bismuth — Tripotassium bismuth dicitrate 300 mg tablet
  Other Names: Denol
  Arms: MTN 500 mg+TCL 500 mg+BIS 300 mg; Tegoprazan 50 mg+MTN 500 mg+TCL 500 mg+BIS 300 mg

SUMMARY:
This study aims to evaluate the pharmacokinetic interaction between tegoprazan and combination of metronidazole, tetracycline and bismuth in healthy adult volunteers.

DETAILED DESCRIPTION:
A open-label, randomized, multiple dose, two arm, two period, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥ 19 and < 55 year-old on the day of obtaining the informed consent.
* Body mass index (BMI) ≥ 17.5 kg/m2 and < 28.0 kg/m2 with a body weight ≥ 55 kg at screening.
* H. pylori negative.

Exclusion Criteria:

* Medical History

  1. History or evidence of clinically significant disease
  2. History of gastrointestinal disease (e.g., esophageal disease such as esophageal achalasia or stenosis, and Crohn's disease) or surgery that may affect the absorption of a drug.
  3. History or presence of hypersensitivity to IMPs, components of IMPs, benzimidazoles, imidazole derivatives or tetracycline antibiotics
* Laboratory tests(in blood)

  1) Total bilirubin, AST (GOT), ALT (GPT) > 1.5 X upper limit of normal (ULN) at screening
* History of drug/alcohol abuse
* Participated in other study and received investigational product within 3 months prior to the first study dose.
* taken a medication known to substantially induce or inhibit a drug metabolizing enzyme
* Not able to use a medically acceptable contraceptive method throughout the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
AUC0-12 of tegaprazan and metabolite M1 | pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in period1 ,2.
  Area under the plasma concentration versus time curve of tegoprazan
Cmax of tegaprazan and metabolite M1 | pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in period1 ,2.
  Peak Plasma Concentration of tegoprazan and metabolite M1
AUC0-6 of metronidazole, tetracycline and bismuth | pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in period1 ,2.
  Area under the plasma concentration versus time curve of metronidazole, tetracycline and bismuth
Cmax of metronidazole, tetracycline and bismuth | pre-dose on Day 1,5,6,7 and post-dose up to 24 hours on Day 7 in period1 ,2.
  Peak Plasma Concentration of metronidazole, tetracycline and bismuth

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, Principal Investigator — Chonbuk university hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

REFERENCES:
- [Derived] Jeon JY, Kim SY, Moon SJ, Oh K, Lee J, Kim B, Song GS, Kim MG. Pharmacokinetic Interactions between Tegoprazan and Metronidazole/Tetracycline/Bismuth and Safety Assessment in Healthy Korean Male Subjects. Clin Ther. 2021 Apr;43(4):722-734. doi: 10.1016/j.clinthera.2021.01.026. Epub 2021 Feb 23. PMID 33637332